CLINICAL TRIAL: NCT03961672
Title: A Phase II Study of Intermittent Duvelisib Dosing in Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Brief Title: Intermittent Duvelisib Dosing in Treating Patients With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19563; NCI-2019-02789 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HEM-19009-LM; 19563 (City of Hope); STUDY00019402 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2019-05-14; First posted 2019-05-23 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — duvelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (duvelisib) (Experimental): INDUCTION: Patients receive duvelisib PO BID on days 1-28. Cycles repeat every 28 days for 12 weeks in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive duvelisib PO BID on days 1-2, 8-9, 15-16, and 22-23. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Duvelisib

INTERVENTIONS:
Drug: Duvelisib — Given PO
  Other Names: 8-Chloro-2-phenyl-3-((1S)-1-(7H-purin-6-ylamino)ethyl)isoquinolin-1(2H)-one; Copiktra; INK-1197; IPI-145

SUMMARY:
This phase II trial studies how well duvelisib on an intermittent (irregular) dosing schedule works in treating patients with chronic lymphocytic leukemia or small lymphocytic lymphoma. Duvelisib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving duvelisib on an intermittent schedule may result in similar effectiveness with less amount of severe side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of duvelisib (induction followed by maintenance [intermittent dosing]) in patients with relapsed or refractory chronic lymphocytic leukemia (CLL), as measured by the progression free survival (PFS).

SECONDARY OBJECTIVES:

I. To evaluate safety of duvelisib induction and maintenance (by intermittent dosing) in relapsed/refractory CLL.

II. To evaluate clinical benefits to duvelisib treatment.

EXPLORATORY OBJECTIVE:

I. To evaluate T-cell populations in patients with CLL treated with duvelisib.

OUTLINE:

INDUCTION: Patients receive duvelisib orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days for 12 weeks in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive duvelisib PO BID on days 1-2, 8-9, 15-16, and 22-23. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Histologically or flow cytometry confirmed diagnosis of B-CLL/small lymphocytic lymphoma (SLL) according to National Cancer Institute - Working Group (NCI-WG) 1996 guidelines. Patients who lack CD23 expression on their leukemia cells should be examined for (and found NOT to have) either t(11;14) or cyclin D1 overexpression, to rule out mantle cell lymphoma.
* Participants have undergone >= 1 prior chemotherapy-based or immunotherapy-based regimen or targeted therapy (e.g., inhibitors of BTK [e.g., ibrutinib], or BCL2 [e.g., venetoclax]) administered for >= 2 cycles (>= 8 weeks for oral therapies), and have had either documented disease progression or no response (i.e., stable disease [SD]) to the most recent treatment regimen.

  * Note: Individuals intolerant to ibrutinib therapy and those who progress on ibrutinib are eligible as long as they satisfy the above criteria.
* Patients with CLL/SLL must demonstrate active disease meeting at least 1 of the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2018 criteria for requiring treatment:

  * A minimum of any one of the following constitutional symptoms:

    * Unintentional weight loss > 10% within the previous 6 months prior to screening.
    * Extreme fatigue (unable to work or perform usual activities).
    * Fevers of greater than 100.5 degrees Fahrenheit (F) for >= 2 weeks without evidence of infection.
    * Night sweats without evidence of infection.
  * Evidence of progressive marrow failure as manifested by the development of, or worsening of anemia or thrombocytopenia.
  * Massive (i.e., > 6 cm below the left costal margin), progressive or symptomatic splenomegaly.
  * Massive nodes or clusters (i.e., > 10 cm in longest diameter) or progressive lymphadenopathy.
  * Progressive lymphocytosis with an increase of > 50% over a 2-month period, or an anticipated doubling time of less than 6 months.
  * Autoimmune anemia or thrombocytopenia that is poorly responsive to corticosteroids.
  * Symptomatic or functional extranodal involvement (eg, skin, kidney, lung, spine)
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status =< 2.
* Direct bilirubin =< 2 x institutional upper limit of normal (ULN); unless due to known Gilbert's syndrome or compensated hemolysis directly attributable to CLL (prior to starting study drug).
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) less than 2.5 x institutional ULN (prior to starting study drug).
* Estimated creatinine clearance (CrCL) using the Cockcroft-Gault equation (or an alternative equation, per institutional standard) >= 30 mL/min (prior to starting study drug).
* Platelets >= 30,000/mm^3 independent of transfusion support, with no active bleeding, and absolute neutrophil count (ANC) >= 500/mm^3, unless due to disease involvement in the bone marrow (prior to starting study drug).
* Participant must be able to swallow tablets or capsules. A participant with any gastrointestinal disease that would impair ability to swallow, retain, or absorb drug is not eligible.
* Female participants of childbearing potential (defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally postmenopausal for at least 12 consecutive months for women > 55 years of age) must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female participants of childbearing potential must agree to use adequate methods of contraception starting with the first dose of study therapy through 60 days after the last dose of study therapy.

  * Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year without an alternative medical cause.
* Male participants must agree to use an adequate method of contraception starting with the first dose of study therapy through 60 days after the last dose of study therapy.

Exclusion Criteria:

* Prior therapeutic intervention with any of the following:

  * Therapeutic anticancer antibodies within 4 weeks;
  * Radio- or toxin-immunoconjugates within 10 weeks;
  * Inhibitors of Bruton tyrosine kinase (BTK) (e.g., ibrutinib), BH3-mimetic venetoclax, lenalidomide and other "targeted" therapy - within 6 half-lives (i.e., 36 hours for ibrutinib)
  * All other chemotherapy, radiation therapy within 3 weeks prior to initiation of therapy.
  * PI3K inhibitors (idelalisib, copanlisib or any investigational PI3K inhibitor including duvelisib and umbralisib) at any time.
* Any adverse event related to prior therapy that has not recovered to grade =< 1.
* Chronic use of corticosteroids in excess of prednisone 30 mg/day or its equivalent.
* Allogeneic stem cell transplant within the past 12 months, or ongoing immunosuppressive therapy other than prednisone =< 10 mg/day (or equivalent).
* Use of strong CYP3A4 inhibitors or inducers, in the one week prior to initiating study treatment or concomitant.
* Unable to receive prophylactic treatment for pneumocystis, herpes simplex virus (HSV), or herpes zoster (varicella zoster virus [VZV]) at screening.
* History of prior malignancy except:

  * Malignancy treated with curative intent and no known active disease present for >= 2 years prior to initiation of therapy on current study;
  * Adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease;
  * Adequately treated in situ carcinomas (e.g., breast, cervical, esophageal, etc.) without evidence of disease;
  * Asymptomatic prostate cancer managed with "watch and wait" strategy
* Uncontrolled immune hemolysis or thrombocytopenia (positive direct antiglobulin test in absence of hemolysis or history of immune-mediated cytopenias are not exclusions).
* History of human immunodeficiency virus (HIV) infection or active hepatitis B or C.
* History of chronic liver disease.
* Major surgery (requiring general anesthesia) within 2 weeks prior to initiation of therapy.
* Patients with clinically significant medical condition of malabsorption, inflammatory bowel disease, chronic conditions which manifest with diarrhea, refractory nausea, vomiting or any other condition that will interfere significantly with drug absorption.
* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or a pacemaker within the last 6 months prior to screening.
* Baseline QT interval corrected with Fridericia's method (QTcF) > 500 ms. (NOTE: criterion does not apply to subjects with a right or left bundle branch block BBB).
* Active uncontrolled infection.
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2026-10-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alexey V Danilov, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - OHSU Knight Cancer Institute, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38836342/

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Duvelisib): INDUCTION: Patients receive duvelisib PO BID on days 1-28. Cycles repeat every 28 days for 12 weeks in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive duvelisib PO BID on days 1-2, 8-9, 15-16, and 22-23. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Duvelisib: Given PO
Period: Overall Study
Arm/Group | Treatment (Duvelisib)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Duvelisib)
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 74 [59 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) at 12 Months
Description: Progression is defined using IWCLL 2018 guidelines (Section 5.3 of Hallek et al, 2018). Proportion of subjects achieving 12-month PFS were estimated along with a two-sided exact Clopper-Pearson 95% confidence interval. PFS was estimated from start of duvelisib treatment until death, time of progression, start of new therapy, or end of follow-up, whichever occurs first. PFS was censored at the start of new therapy or end of follow-up, whichever occurs first.
Time Frame: First dose of duvelisib until death, time of progression, start of new therapy, or 12 months from start of therapy, whichever occurs first
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Duvelisib)
Number analyzed (Participants) | 15
percentage of participants | 48 [21 to 71]

2. Secondary Outcome: Objective Response Rate (ORR) (Including Complete Response [CR] and Partial Response [PR])
Description: Treatment responses were defined by using IWCLL 2018 guidelines (Hallek et al, 2018). Overall Response (OR) = CR + PR. Probability of having ORR was measured and reported with 95% exact confidence interval.
Time Frame: First dose of duvelisib up to 12 months after discontinuation of duvelisib
Population: 4 participants were not evaluated for response due to early discontinuations for toxicity, myelodysplastic syndrome and COVID-19.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Duvelisib)
Number analyzed (Participants) | 11
percentage of participants | 82 [48 to 98]

3. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: Progression is defined using IWCLL 2018 guidelines (Section 5.3 of Hallek et al, 2018). Estimated distribution of the PFS was plotted using Kaplan Meier curves and reported with median PFS and 95% confidence intervals.
Time Frame: First dose of duvelisib until death, time of progression, or start of new therapy, whichever occurs first, assessed up to 12 months after discontinuation of duvelisib
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Duvelisib)
Number analyzed (Participants) | 15
months | 9.9 [5.5 to 29]

4. Secondary Outcome: Percentage of the Participants With 12-month Duration of Response (DOR)
Description: Duration of response (DOR), for participants who responded to the study intervention, was measured from the time of first documented objective response (i.e., CR or PR/PR-L) until evidence of progressive disease, start of new therapy, death, or end of follow-up. DOR was censored at the start of new therapy or end of follow-up, whichever occurs first. Proportion of the participants achieving 12-month DOR and the 95% confidence interval were reported.
Time Frame: From time of ORR until death, time of progression, start of new therapy, or end of follow-up, whichever occurs first, assessed up to 12 months after discontinuation of duvelisib
Population: 9 participants achieved objective responses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Duvelisib)
Number analyzed (Participants) | 9
percentage of participants | 30 [5 to 61]

5. Secondary Outcome: Percentage of Participants With Grade 3 4 5 Toxicity Related to Duvelisib
Description: Percentage of participants, that received at least one dose of duvelisib, had developed grade 3 4 5 toxicities at least possibly related to duvelisib. The 95% confidence interval was calculated by the Clopper-Pearson (exact) method.
Time Frame: From first dose of duvelisib until 3 months post-discontinuation of duvelisib
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Duvelisib)
Number analyzed (Participants) | 15
percentage of participants | 67 [38 to 88]

6. Secondary Outcome: Number of Administrated Cycles of the Study Treatment
Description: Number of study treatment cycles that participants received from the first dose of study drug until therapy was discontinued for any reason.
Time Frame: From first dose of duvelisib until time of duvelisib discontinuation up to 5 years.
Measure: Median (Full Range); unit: cycles
Arm/Group | Treatment (Duvelisib)
Number analyzed (Participants) | 15
cycles | 5 [1 to 31]

ADVERSE EVENTS:
Time Frame: Averse events were assessed from the initial treatment to 30 calendar days after the last study drug dose. Adverse events were monitored and assessed at each cycle of the study treatment. Vital status was assessed from the initial treatment up to 12 months after the end of the treatment.
Arm/Group | Treatment (Duvelisib)
All-Cause Mortality (participants affected / at risk) | 3/15
Serious Adverse Events (participants affected / at risk) | 7/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Duvelisib) (N=15)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
HEART FAILURE (Cardiac disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
SCC TUMOR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Duvelisib) (N=15)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 4 (5)
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 2 (2)
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (3)
HEART FAILURE (Cardiac disorders) | 1 (1)
PALPITATIONS (Cardiac disorders) | 2 (2)
SINUS TACHYCARDIA (Cardiac disorders) | 2 (2)
RIGHT EYE RED (Eye disorders) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3)
COLITIS (Gastrointestinal disorders) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 5 (13)
ESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 2 (8)
NAUSEA (Gastrointestinal disorders) | 5 (6)
PANNICULTIS (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 5 (6)
BODY ACHES (General disorders) | 1 (1)
CERVICAL LYMPH NODE SWELLING FROM BUG BITE ON NECK (General disorders) | 1 (1)
CHILLS (General disorders) | 4 (5)
FATIGUE (General disorders) | 8 (9)
FEVER (General disorders) | 1 (3)
FLU LIKE SYMPTOMS (General disorders) | 1 (1)
GAIT DISTURBANCE (General disorders) | 1 (1)
PAIN (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (2)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
BRUISING (Injury, poisoning and procedural complications) | 2 (2)
FALL (Injury, poisoning and procedural complications) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 (16)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 4 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (15)
BLOOD BILIRUBIN INCREASED (Investigations) | 2 (3)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 4 (6)
CREATININE INCREASED (Investigations) | 2 (3)
LYMPHOCYTE COUNT INCREASED (Investigations) | 4 (4)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 (3)
PLATELET COUNT DECREASED (Investigations) | 5 (10)
WEIGHT LOSS (Investigations) | 2 (2)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERKALEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERURICEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 2 (3)
HYPONATREMIA (Metabolism and nutrition disorders) | 2 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
COMPRESSION FRACTURE (T9) (Musculoskeletal and connective tissue disorders) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 2 (2)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (2)
HEADACHE (Nervous system disorders) | 5 (5)
NEUROPATHY "INTERMITTENT ELECTRICAL SHOCKS TO FEET/LOWER LEGS" (Nervous system disorders) | 1 (1)
PARESTHESIA (Nervous system disorders) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (2)
ANXIETY (Psychiatric disorders) | 1 (1)
CONFUSION (Psychiatric disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PRURITIC RASH ON ARMS (Skin and subcutaneous tissue disorders) | 1 (1)
SPOT ON HEAD (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1)
FLUSHING (Vascular disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 4 (8)
HYPOTENSION (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT03961672/Prot_SAP_000.pdf